CLINICAL TRIAL: NCT05180448
Title: Sharing Digital Self-Monitoring Data With Others to Enhance Long-Term Weight Loss: A Randomized Trial Using a Factorial Design
Brief Title: Sharing Digital Self-Monitoring Data With Others to Enhance Long-Term Weight Loss
Acronym: FitLink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R01DK129300 (NIH); 1R01DK129300-01 (NIH)
Record Dates: First submitted 2021-09-20; First posted 2022-01-06 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Overweight; Obesity
Keywords: weight loss; lifestyle modification; behavioral modification; overweight; obesity
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: This is a 2x2x2 design. There are three factors, each with two levels: ON vs OFF
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blind to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Coach Share On + Group Share On + Friend/Family Share On (Experimental)
  Interventions: Behavioral: Coach Share On; Behavioral: Group Share On; Behavioral: Friend/Family Share On; Behavioral: Behavioral Weight Loss Treatment
- Coach Share On + Group Share On + Friend/Family Share Off (Experimental)
  Interventions: Behavioral: Coach Share On; Behavioral: Group Share On; Behavioral: Friend/Family Share Off; Behavioral: Behavioral Weight Loss Treatment
- Coach Share On + Group Share Off + Friend/Family Share On (Experimental)
  Interventions: Behavioral: Coach Share On; Behavioral: Friend/Family Share On; Behavioral: Group Share Off; Behavioral: Behavioral Weight Loss Treatment
- Coach Share On + Group Share Off + Group Share Off (Experimental)
  Interventions: Behavioral: Coach Share On; Behavioral: Group Share Off; Behavioral: Friend/Family Share Off; Behavioral: Behavioral Weight Loss Treatment
- Coach Share Off + Group Share On + Friend/Family Share On (Experimental)
  Interventions: Behavioral: Group Share On; Behavioral: Friend/Family Share On; Behavioral: Coach Share Off; Behavioral: Behavioral Weight Loss Treatment
- Coach Share Off + Group Share On + Friend/Family Share Off (Experimental)
  Interventions: Behavioral: Group Share On; Behavioral: Coach Share Off; Behavioral: Friend/Family Share Off; Behavioral: Behavioral Weight Loss Treatment
- Coach Share Off + Group Share Off + Friend/Family Share On (Experimental)
  Interventions: Behavioral: Friend/Family Share On; Behavioral: Coach Share Off; Behavioral: Group Share Off; Behavioral: Behavioral Weight Loss Treatment
- Coach Share Off + Group Share Off + Friend/Family Share Off (Experimental)
  Interventions: Behavioral: Coach Share Off; Behavioral: Group Share Off; Behavioral: Friend/Family Share Off; Behavioral: Behavioral Weight Loss Treatment

INTERVENTIONS:
Behavioral: Coach Share On — If an index participant is randomized to have Coach Share ON, the coach will have continuous access to objective, real-time, detailed device data, and address data directly in all individual interactions with index participants (groups, individual weigh-ins, phone calls, texts), conveying that they are closely monitoring progress.
  Arms: Coach Share On + Group Share Off + Friend/Family Share On; Coach Share On + Group Share Off + Group Share Off; Coach Share On + Group Share On + Friend/Family Share Off; Coach Share On + Group Share On + Friend/Family Share On
Behavioral: Group Share On — If Group Share is ON, participants in a given LM group will view and respond to aspects of each other's self-monitoring device data in their small-group text messages. Each small group participant's data will be highlighted one day of the month, and content from the Group Share Off message library also will be sent.
  Arms: Coach Share Off + Group Share On + Friend/Family Share Off; Coach Share Off + Group Share On + Friend/Family Share On; Coach Share On + Group Share On + Friend/Family Share Off; Coach Share On + Group Share On + Friend/Family Share On
Behavioral: Friend/Family Share On — Index participants who are randomized to have Friend/Family Share ON will give their friend or family member access to their self-monitoring data. Text messages sent by the program bot, which includes the index participant and friend/family member, will use a similar format as described in Group Share ON. The friend or family member will be trained to respond to data in ways that enhance the participant's motivation and self-regulation.
  Arms: Coach Share Off + Group Share Off + Friend/Family Share On; Coach Share Off + Group Share On + Friend/Family Share On; Coach Share On + Group Share Off + Friend/Family Share On; Coach Share On + Group Share On + Friend/Family Share On
Behavioral: Coach Share Off — Among index participants who are randomized to have Coach Share OFF, the coach will have no access to their device data. Index participants will be explicitly told their coach does not have data access. During groups and phone calls, the participant will self-report progress, and goal setting will be based on that self-report. Text messages from the coach will be personalized in the OFF condition, as they are when coach data sharing is ON, though these messages will not be informed by device data. Instead, text messages will provide a reminder of key goals and strategies discussed in the previous phone call and provide encouragement for participant efforts.
  Arms: Coach Share Off + Group Share Off + Friend/Family Share Off; Coach Share Off + Group Share Off + Friend/Family Share On; Coach Share Off + Group Share On + Friend/Family Share Off; Coach Share Off + Group Share On + Friend/Family Share On
Behavioral: Group Share Off — Among index participants randomized to have Group Share OFF, supportive accountability will not be the target of participant interactions and no data will be shared with LM program peers. Instead, once weekly prompts for small group text exchanges will encourage index participants to provide social support (primarily of the informational type) to each other. Index participants will be explicitly told that they should not include information on goal progress such as weight change or minutes of PA.
  Arms: Coach Share Off + Group Share Off + Friend/Family Share Off; Coach Share Off + Group Share Off + Friend/Family Share On; Coach Share On + Group Share Off + Friend/Family Share On; Coach Share On + Group Share Off + Group Share Off
Behavioral: Friend/Family Share Off — If an index participant is randomized to Friend/Family Share OFF, the text messages from the bot will prompt the participant and friend/family member to communicate about the LM program; those messages will be standardized, except for names, and will not be tailored to index participant progress. Index participants will be instructed to refrain from sharing any device data with friends or family members.
  Arms: Coach Share Off + Group Share Off + Friend/Family Share Off; Coach Share Off + Group Share On + Friend/Family Share Off; Coach Share On + Group Share Off + Group Share Off; Coach Share On + Group Share On + Friend/Family Share Off
Behavioral: Behavioral Weight Loss Treatment — Standard Behavioral Weight Loss Treatment (remotely delivered)

SUMMARY:
Adults attempting weight loss through lifestyle modification (LM) typically find maintenance of behavior change difficult. Outcomes might be improved if participants are provided with sustained sources of accountability and support and ongoing opportunities to reflect with others on goal progress. This study proposes that sharing digital data with other parties has the potential to improve long-term weight loss. The proposed study will enroll adults ("index participants") (N = 320) with overweight/obesity in a 24-month LM program and instruct them to use digital tools for self-monitoring of weight, physical activity, and eating on a daily basis.

DETAILED DESCRIPTION:
Adults attempting weight loss through lifestyle modification (LM) typically find maintenance of behavior change difficult. Outcomes might be improved if participants are provided with sustained sources of accountability and support and ongoing opportunities to reflect with others on goal progress. This study proposes that sharing digital data with other parties has the potential to improve long-term weight loss. The proposed study will enroll adults ("index participants") (N = 320) with overweight/obesity in a 24-month LM program and instruct them to use digital tools for self-monitoring of weight, physical activity, and eating on a daily basis. Groups will meet remotely each week in months 1-3 to initiate weight loss. In months 4-24, intervention contact will be remote and will include the following: quarterly group meetings held via videoconference; brief phone calls with the coach held twice per quarter; and monthly text messages with the coach, with a small group of fellow group participants, and with a friend or family member outside of the program. Text message content will vary according to treatment condition, i.e. three types of data sharing partnerships: Coach Share, Group Share, and Friend/Family Share. Outcomes will be measured at months 0, 3, 6, 12, and 24. Primary aims include determining if Coach Share, Group Share, and Friend/ Family Share each improve long-term weight loss, PA, and calorie intake, and examining if effects are additive when participants are assigned to engage in more than one type of data sharing partnership. The secondary aim is to explore mediators and moderators of intervention effects. The tertiary aim is to determine how the quality of relationship with coach, group members, and friends/family member over time may differentially moderate treatment effects and predict data sharing efficacy. As digital technology makes data sharing increasingly feasible, it is critical to determine how to optimize these partnerships to improve long-term outcomes in LM.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be of overweight or obese BMI (27-50 kg/m2)
* Individuals must be adults (aged 18-70)
* Able to engage in physical activity (defined as walking two city blocks without stopping)
* Access and willingness to use a smartphone and internet
* Has one adult friend or family member who indicates willingness to serve in a support role
* Satisfactory completion of all enrollment procedures
* English Speaking

Exclusion Criteria:

* Medical or psychiatric condition (e.g., cancer, type I diabetes, psychosis, full-threshold eating disorder) that may pose a risk to the participant during intervention or cause a change in weight, or limit ability to comply with the program or participate appropriately in group-based treatment
* Currently pregnant or breastfeeding, or planning to become pregnant in the next 24 months
* Use of insulin or a medication that can cause significant change in weight
* History of bariatric surgery
* Weight loss of greater than or equal to 5% in the previous 3 months
* Weight loss of greater than or equal to 10% in the past 3 years that is currently being maintained

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Weight | 0 month, 3 month, 6 month, 12 month, 24 month
  Weight will be measured using a wireless scale. In order to maximize accuracy, we will (1) provide instructions (e.g., place scale on flat, hard surface; weigh upon waking, without clothes, after using the bathroom), (2) require participants to confirm that they are following instructions at each assessment point, (3) remove errant weights (e.g., >1 kg change in 1 day).

SECONDARY OUTCOMES:
Physical Activity | 0 month, 3 month, 6 month, 12 month, 24 month
  Minutes per week of moderate-to-vigorous PA will be measured by using FitBit. Steps per day from the Fitbit also will be examined.
Calorie Intake | 0 month, 3 month, 6 month, 12 month, 24 month
  Average calorie intake over 7 days will be derived from the Fitbit digital food log as a secondary outcome.

OTHER OUTCOMES:
Perceived Supportive Accountability for Weight Control | 0 months, 6 month, 12 month, 24 month
  (mediator, moderator) will be measured with the Supportive Accountability Measure and the Supportive Accountability Inventory
Self-regulation value of program components | 3 months, 6 month, 12 month, 24 month
  (Mediator, moderator) will be measured with items, adapted from previous research, that ask index participants to rate how helpful each program component is reflecting on how their progress compares to their goals, planning short-term behaviors and strategy use, and evaluating if current goals should be adjusted.
Self-monitoring | Calculated continuously for 24 months
  (Mediator, moderator) will be objectively measured as the number of days in which digital devices were used to measure weight, record eating, or PA.
social comparison | 0, 12, 24 months
  (Mediator, moderator) will be measured with the Iowa-Netherlands Comparison Orientation Measure, with items modified to be focused on the lifestyle modification group.
Perceived Social Support | 0 months, 6 month, 12 month, 24 month
  (Mediator, moderator) assessed with the Social Support for Healthy Behaviors Measure. Index participants will report the frequency with which friends and family members engaged in behaviors that support or undermine healthy eating and physical activity in the past month.
Relationship Quality | 0, 3, 6, 12, 24 months
  (Moderator, moderator) will be measured with items adapted from the client version of the Working Alliance Inventory-Bond Subscale. Ratings will be completed separately for the relationship with the coach, the lifestyle modification group, and the designated friend/family support person, yielding scores for each party
Weight Self-Stigma | 0 months
  (moderator) will be measured with items, adapted from previous research, that assess for weight self-stigma.
Friend/family characteristics | 0, 3, 6, 12, 24 months
  (mediator, moderator) Items to characterize the friend/family member relationship, such as their age, gender, body size, perceived healthfulness of diet, interest in weight loss, frequency of communication, comfort discussion lifestyle modification with them, reactions to weight-related communication
Small group dynamic | 3, 6, 12, 24 months
  (mediator, moderator) Items to characterize the small group dynamic, including frequency of communication and reactions to communication
Demographic variables | 0 months
  (moderator) Items to characterize the participant, including age, sex, race, ethnicity, education level, household composition
Coach characteristics | 0 months
  (moderator) Coach level of behavioral weight loss experience (# of sessions previously conducted) and level of education will be calculated
Method of message delivery | 0 months
  (moderator) Whether text messages were delivered to app (Wave 1 and 2) or via SMS (Wave 3 and 4) will be examined to determine if this impacts intervention efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Meghan L Butryn, PhD, Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/48/NCT05180448/Prot_ICF_001.pdf